CLINICAL TRIAL: NCT03245983
Title: Spirituality, Experience of Disease and Quality of Life in Cancer Patients
Acronym: SPIQOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-32
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Psychology and Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient willing to participate (Experimental)
  Interventions: Behavioral: Questionnaire and interview

INTERVENTIONS:
Behavioral: Questionnaire and interview — Cancer patients will answer questionnaires and will be interviewed by a pshychologist to assess their spirituality and quality of life toward their disease

SUMMARY:
The general aim of research is to identify and analyze the impact and role of spirituality (as a search for meaning and understanding of the meaning of existence) in the experience of cancer. For this purpose, the main objective of this study is to measure the "existential" component in the trajectory of the disease. It is a question of observing its potential contribution to the improvement of the quality of life of the patients and to define if this variable can be translated into a strategy of adjustment for the patients. This research has a double interest: (a) clinical interest in better managing patients' needs; (B) an interest in research in the field of health by combining a measure of spirituality with other psycho-social variables.

The project is a prospective non-randomized mono-centric study by questionnaire and research interview. It is a study that seeks to identify the role of spirituality in the experience of illness (i.e. representations, adjustments, emotional distress) and as a determinant of the quality of life of subjects with cancer pathology.

The interviews will be conducted by a psychologist to qualitatively collect the elements of the lived experience of the disease in connection with the spiritual elements of the "quest for meaning" type.

The population covered by the project is in and out patients coming to the Department of Medical Oncology and Palliative Care at the CHU de la Timone.

The realization of this project will allow investigators to explore the specificity of the existential / spiritual dimensions of patients confronted with cancer, to assess the patients' needs for this type of approach within the hospital, to link the existential component / Spiritual with psycho-social variables

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing chemotherapy

Exclusion Criteria:

* patient presenting psychiatric or neurological disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of quality of life in patient cancer | 36 months
  Questionnaires(QLQC30) for patients with cancer.
Descriptive analysis of spirituality role in cancer patient | 36 month
  Spirituality Index of Well-Being questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique -Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided